CLINICAL TRIAL: NCT02769052
Title: Transcutaneous Electrical Nerve Stimulation (TENS) Self-applied as Complementary Treatment for Pain and Its Impact on Quality of Life and Sexuality of Women With Deep Endometriosis: Randomized Controlled Trial
Brief Title: TENS Self-applied in the Complementary Treatment of Deep Endometriosis
Acronym: tici_mira
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Ticiana Aparecida Alves de Mira, PhD, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 51799115.3.1001.5404
Record Dates: First submitted 2016-05-06; First posted 2016-05-11 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Endometriosis
Keywords: endometriosis; dyspareunia; physical therapy; sexuality; transcutaneous electrical nerve stimulation
MeSH Terms: conditions — Endometriosis; Dyspareunia; Sexuality | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Follow-up/Treatment - Control Group (Active Comparator): Composed of two phases of 8 weeks each (follow-up - treatment). The treatment using the self-applied Transcutaneous Electrical Nerve Stimulation (TENS) will prescribe with daily application, twice a day for 20 minutes each application.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- Treatment Group (Active Comparator): Composed of one phase of 8 weeks (treatment). The treatment using the self-applied Transcutaneous Electrical Nerve Stimulation (TENS) will prescribe with daily application, twice a day for 20 minutes each application.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — Electrotherapy through self-applied device .

SUMMARY:
Objective: to evaluate the effectiveness of Transcutaneous Electrical Nerve Stimulation (TENS) self-applied for the treatment of pain and the impact of this therapy on quality of life and sexuality of women with deep endometriosis.

DETAILED DESCRIPTION:
* Women will be selected to participate in the study between June 2016 to March 2018, from medical records research and routine queries in Endometriosis clinic of the Gynecology's Hospital of University of Campinas (UNICAMP) and the clinic of Gynecology (Endometriosis routine queries) of the Hospital of University of São Paulo (USP). All women will respond to the Check List for inclusion in the study and will sign an informed consent form.
* The women selected will be randomized into two distinct groups: follow-up/treatment - control group (CG) composed of two phases of 8 weeks each or treatment group (TG) consists of one phase of 8 weeks. The randomization will be through sealed brown envelopes, whose numerical sequence will be generated by computer programming in Statistical Analysis System (SAS), held by a person not participating in the study. Once allocated, all women respond to a clinical and socio-demographic questionnaire, Visual analog scale; Deep Dyspareunia scale; Diagram of Location and characterization of Pain; Endometriosis Health Profile (EHP-30); Female Sexual Function Index pre-and post-treatment. In addition, the woman will fill a daily control of pain.

All procedures of the study will be carried out by the same researcher, to enforce the search protocol. After the end of the collection, all data will be entered in the Excel program for Windows and conferred for a second digitizer.

* The sample size calculation was based on the pilot study developed by Mira et al. (2015) whereas the use of the TENS for relief of chronic pelvic pain and deep dyspareunia generated by endometriosis, whose pre-and post-treatment discomfort was assessed by Visual analog scale (EVA). The number of women in this study was of 22 women divided into two treatment groups. Applied for the calculation of sample size, the t test for independent variables to the study cited and given a power of test 90% and significance level of 5%, the sample size obtained was of 24 patients in total. Considering the following loss of 20%, the total number shall be 29 women, divided into two groups: follow-up/treatment group (n = 15) and treatment/monitoring group (n = 14). For better quantification of all the variables involved, we will seek ideally a total of 80 women, divided into two groups (n = 40).
* The data obtained will be described by mean ± standard deviation. The results will be tested for normal distribution using the Shapiro-Wilk test. For analysis of the second sample groups, features will be used the Fisher exact test. For comparison of means obtained from scales and questionnaires, pre-and post-intervention, t-test will be used or non-parametric analog, for each variable, previously cited. The comparison of variables between groups will be analyzed by t test or nonparametric analog. Significance will be considered through the value p <.05. The data will be analyzed by intention to treat. The software used for statistical analysis SAS version 9.2.

ELIGIBILITY:
Inclusion Criteria:

* Women at reproductive age;
* 18 and 50 years;
* diagnosis of deep endometriosis (cul-de-sac and intestinal lesions);
* using hormonal treatment at least 3 months;
* persistence of chronic pelvic pain and/or dyspareunia.

Exclusion Criteria:

* Women with decreased skin sensitivity;
* pregnant women;
* women with pacemaker implants;
* cutaneous hypersensitivity (allergic reactions to gel or electrode);
* women with epilepsy;
* cardiac (cardiac arrhythmia);
* osteosynthesis in the application place;
* a solution of discontinuity of the skin;
* malignant tumors;
* acute inflammatory disease;
* other gynecological associated pathologies;
* a cognitive deficiency that precludes the understanding of instruments and/or instructions for self-applied of TENS.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-06; Primary Completion 2018-03 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Improvement of Pelvic Pain | up to one year
  The chronic pelvic pain will be evaluated by specific instrument (Visual Analogue Scale).
Improvement of Pain during the relation | up to one year
  The deep dyspareunia will be evaluated by specific instrument (Deep Dyspareunia Scale).

SECONDARY OUTCOMES:
Improvement of Quality of life | up to one year
  The quality of life will be accessed by one specific questionnaire for endometriosis.
Improvement of Sexuality | up to one year
  The sexuality will be accessed by questionnaire.
Improvement of The global pain | up to one year
  The global pain will be evaluated by Diagram Localization and Characterization of Pain (design body representation).

CONTACTS AND LOCATIONS:
Overall Officials: Ticiana AA Mira, MSc, Principal Investigator — University of Campinas; Cristina L Benetti-Pinto, PhD, Study Chair — University of Campinas
Locations (1):
- Gynecology Hospital, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dizerega GS, Barber DL, Hodgen GD. Endometriosis: role of ovarian steroids in initiation, maintenance, and suppression. Fertil Steril. 1980 Jun;33(6):649-53. doi: 10.1016/s0015-0282(16)44780-1. PMID 6769717
- [Background] Kennedy S, Bergqvist A, Chapron C, D'Hooghe T, Dunselman G, Greb R, Hummelshoj L, Prentice A, Saridogan E; ESHRE Special Interest Group for Endometriosis and Endometrium Guideline Development Group. ESHRE guideline for the diagnosis and treatment of endometriosis. Hum Reprod. 2005 Oct;20(10):2698-704. doi: 10.1093/humrep/dei135. Epub 2005 Jun 24. PMID 15980014
- [Background] Ferrero S, Esposito F, Abbamonte LH, Anserini P, Remorgida V, Ragni N. Quality of sex life in women with endometriosis and deep dyspareunia. Fertil Steril. 2005 Mar;83(3):573-9. doi: 10.1016/j.fertnstert.2004.07.973. PMID 15749483
- [Background] Chwalisz K, Brenner RM, Fuhrmann UU, Hess-Stumpp H, Elger W. Antiproliferative effects of progesterone antagonists and progesterone receptor modulators on the endometrium. Steroids. 2000 Oct-Nov;65(10-11):741-51. doi: 10.1016/s0039-128x(00)00190-2. PMID 11108885
- [Background] Carpenter SE, Tjaden B, Rock JA, Kimball A. The effect of regular exercise on women receiving danazol for treatment of endometriosis. Int J Gynaecol Obstet. 1995 Jun;49(3):299-304. doi: 10.1016/0020-7292(95)02359-k. PMID 9764869
- [Background] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Background] Scott J, Huskisson EC. Graphic representation of pain. Pain. 1976 Jun;2(2):175-84. No abstract available. PMID 1026900
- [Background] Jones G, Kennedy S, Barnard A, Wong J, Jenkinson C. Development of an endometriosis quality-of-life instrument: The Endometriosis Health Profile-30. Obstet Gynecol. 2001 Aug;98(2):258-64. doi: 10.1016/s0029-7844(01)01433-8. PMID 11506842
- [Background] Mengarda CV, Passos EP, Picon P, Costa AF, Picon PD. [Validation of Brazilian Portuguese version of quality of life questionnaire for women with endometriosis (Endometriosis Health Profile Questionnaire--EHP-30)]. Rev Bras Ginecol Obstet. 2008 Aug;30(8):384-92. doi: 10.1590/s0100-72032008000800003. Portuguese. PMID 19142521
- [Background] Minson FP, Abrao MS, Sarda Junior J, Kraychete DC, Podgaec S, Assis FD. [Importance of quality of life assessment in patients with endometriosis]. Rev Bras Ginecol Obstet. 2012 Jan;34(1):11-5. Portuguese. PMID 22358342
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451